CLINICAL TRIAL: NCT00536120
Title: A Randomized, Open-Label Study to Assess the Effects of Tysabri Treatment on Vaccination Response and Lymphocyte Subsets in Subjects With Relapsing Forms of Multiple Sclerosis
Brief Title: The Effects of Tysabri Treatment on Vaccination Response and Lymphocyte Subsets in Subjects With Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 101MS404
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Multiple Sclerosis
Keywords: MS; Multiple sclerosis; Relapsing forms of Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab; keyhole-limpet hemocyanin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tysabri Plus Vaccinations (Experimental): Participants receive 9 monthly doses of Tysabri 300 mg intravenous (IV), and receive vaccinations with neoantigen and recall antigen (keyhole limpet hemocyanin [KLH] and tetanus diphtheria toxoid [Td], according to manufacturer's prescribing information) at Month 6 (following the 7th dose of Tysabri) for both KLH and Td, and 14 and 28 days later for KLH.
  Interventions: Biological: BG00002 (natalizumab); Biological: keyhole limpet hemocyanin (KLH); Biological: tetanus diphtheria toxoid vaccine (Td)
- Vaccinations Only (Other): Participants receive only vaccinations with neoantigen and recall antigen (KLH and Td, according to manufacturer's prescribing information) at Month 0 for both KLH and Td, and 14 and 28 days later for KLH. They do not receive any treatment for their MS and remain in the study through Month 2.
  Interventions: Biological: keyhole limpet hemocyanin (KLH); Biological: tetanus diphtheria toxoid vaccine (Td)

INTERVENTIONS:
Biological: BG00002 (natalizumab)
  Other Names: Tysabri
  Arms: Tysabri Plus Vaccinations
Biological: keyhole limpet hemocyanin (KLH) — KLH 1 mg administered subcutaneously (SC) in accordance with the Immucothel investigator's brochure.
  Other Names: Immucothel
Biological: tetanus diphtheria toxoid vaccine (Td) — Td administered in accordance with the manufacturer's prescribing information.

SUMMARY:
The primary objectives of this study were: to evaluate the effect of Tysabri® (natalizumab) on antibody responses after immunization with a neoantigen (keyhole limpet hemocyanin [KLH]) and a recall antigen (tetanus toxoid [Td]), and to evaluate the effect of Tysabri on circulating lymphocyte subsets (CD3+, CD4+, CD8+, CD19+, and CD56+) over time in participants with relapsing forms of multiple sclerosis (MS). The secondary objective was to assess alpha4-integrin saturation and alpha4-integrin expression levels over time.

ELIGIBILITY:
Inclusion Criteria:

* able to give written informed consent
* diagnosis of a relapsing form of MS and must fall within the therapeutic indication stated in the approved label for Tysabri
* aged 18-60 years, inclusive at the time of consent
* free of signs and symptoms suggestive of any serious opportunistic infection, based on medical history, physical examination, or laboratory testing
* must have a known history of tetanus toxoid immunization

Major Exclusion Criteria:

* tetanus toxoid vaccination less than 2 years prior to Screening
* known hypersensitivity to tetanus-diphtheria vaccine or KLH or any other administered vaccinations or their components (such as thimerosal)
* known allergy to shellfish
* history of active tuberculosis or undergoing treatment for tuberculosis
* previous exposure to KLH or vaccines containing KLH components (e.g., cancer vaccines)
* known history of human immunodeficiency virus (HIV), hepatitis C, or hepatitis B infection
* history of, or available abnormal laboratory results indicative of any significant disease
* history of malignancy
* history of organ transplantation (including anti-rejection therapy)
* history of severe allergic or anaphylactic reactions or known drug hypersensitivity
* a clinically significant infectious illness within 30 days prior to the Screening visit
* prior exposure to Tysabri, rituximab, any murine protein, or any therapeutic monoclonal antibody at any time
* receipt of intravenous (IV) or intramuscular (IM) immunoglobulin within 6 months of screening
* live virus, bacterial vaccines, or any other vaccines within 3 months of screening
* treatment with immunosuppressant medications within 6 months prior to screening
* treatment with cyclophosphamide within 1 year prior to screening
* treatment with immunomodulatory medications (interferon beta and glatiramer acetate) within 2 weeks prior to screening
* treatment with systemic corticosteroids within 4 weeks prior to screening
* treatment with any investigational product or approved therapy or vaccination for investigational use within 6 months prior to Screening
* women who are breastfeeding, pregnant, or planning to become pregnant during the study
* female subjects who are not postmenopausal for at least 1 year, surgically sterile (does not include tubal ligation), or willing to practice effective contraception during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (10):
- United States (10):
  - Research Site 1, Fullerton, California
  - Research Site, Centennial, Colorado
  - Research site, Farmington Hills, Michigan
  - Research Site, Patchogue, New York
  - Research Site 3, Charlotte, North Carolina
  - Research Site 5, Oklahoma City, Oklahoma
  - Research Site, Franklin, Tennessee
  - Research Site, Dallas, Texas
  - Research Site 2, Seattle, Washington
  - Research Site 4, Charleston, West Virginia

REFERENCES:
- [Background] Kaufman M, Pardo G, Rossman H, Sweetser MT, Forrestal F, Duda P. Natalizumab treatment shows no clinically meaningful effects on immunization responses in patients with relapsing-remitting multiple sclerosis. J Neurol Sci. 2014 Jun 15;341(1-2):22-7. doi: 10.1016/j.jns.2014.03.035. Epub 2014 Mar 26. PMID 24731783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 10 investigational sites in the US. Study enrollment began on 07 January 2008.
Groups:
- Tysabri Plus Vaccinations: Participants received 9 monthly doses of Tysabri 300 mg intravenous (IV), and received vaccinations with neoantigen and recall antigen (keyhole limpet hemocyanin [KLH] and tetanus diphtheria toxoid [Td], according to manufacturer's prescribing information) at Month 6 (following the 7th dose of Tysabri) for both KLH and Td, and 14 and 28 days later for KLH.
- Vaccinations Only: Participants received only vaccinations with neoantigen and recall antigen (KLH and Td, according to manufacturer's prescribing information) at Month 0 for both KLH and Td, and 14 and 28 days later for KLH. They did not receive any treatment for their MS and remained in the study through Month 2.
Period: Overall Study
Arm/Group | Tysabri Plus Vaccinations | Vaccinations Only
Started | 30 | 30
Completed | 24 | 27
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Positive for Anti-natalizumab Antibodies | 3 | 0
Not completed — Non-compliance | 1 | 0
Not completed — Sponsor Decision Due to Lab Values | 1 | 0
Not completed — Steroid Use | 0 | 2
Not completed — Missed Study Visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tysabri Plus Vaccinations | Vaccinations Only | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (8.34) | 40.4 (9.86) | 41.8 (9.16)
Gender [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 7 | 2 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 29 | 59
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Black or African American | 1 | 4 | 5
  White | 27 | 26 | 53
Time Since First MS Symptoms [Median (Full Range); unit: years] | 8.0 [2 to 31] | 8.5 [2 to 25] | 8.0 [2 to 31]
Time Since First MS Diagnosis [Median (Full Range); unit: years] | 6.0 [1 to 29] | 5.0 [1 to 19] | 5.5 [1 to 29]
Number of Relapses in 3 Years Prior to Screening [Mean (Standard Deviation); unit: relapses] | 3.0 (2.65) | 2.4 (1.83) | 2.7 (2.27)
Number of Relapses in 12 Months Prior to Screening [Mean (Standard Deviation); unit: relapses] | 1.4 (1.07) | 1.0 (0.85) | 1.2 (0.98)
Expanded Disability Status Scale at Screening [Median (Full Range); unit: scores on a scale] — The Expanded Disability Status Scale (EDSS) measures physical disability on a scale from 0.0 (no disability) to 10.0 (death due to disability) in 0.5-point increments.
  scores on a scale | 2.75 [1.0 to 6.0] | 3.00 [0.0 to 7.0] | 3.00 [0.0 to 7.0]
Circulating Lymphocyte Subsets [Mean (Standard Deviation); unit: lymphocyte count/µL] — Circulating lymphocyte subsets (CD3+, CD4+, CD8+, CD19+, and CD56+) at Baseline
  lymphocyte count/µL
    CD3+; n=24 | 1261.5 (309.47) | NA (NA) — Calculated for Tysabri arm only. | 1261.5 (309.47)
    CD4+; n=24 | 905.2 (299.51) | NA (NA) — Calculated for Tysabri arm only. | 905.2 (299.51)
    CD8+; n=24 | 344.6 (123.91) | NA (NA) — Calculated for Tysabri arm only. | 344.6 (123.91)
    CD16+; n=24 | 179.2 (106.12) | NA (NA) — Calculated for Tysabri arm only. | 179.2 (106.12)
    CD19+; n=24 | 269.8 (123.00) | NA (NA) — Calculated for Tysabri arm only. | 269.8 (123.00)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Keyhole Limpet Hemocyanin (KLH) Responders at Day 28 Post-Vaccination
Description: KLH responders were defined as those participants who had at least a 2-fold increase over pre-immunization level of anti-KLH antibodies in their blood at 28 days after vaccination with KLH.
Time Frame: 28 days after immunization (Day 28 for Vaccinations Only Group/Day 196 for Tysabri Plus Vaccinations Group)
Population: Participants with an assessment at Day 28. No imputation methods were used in the primary analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Tysabri Plus Vaccinations | Vaccinations Only
Number analyzed (Participants) | 19 | 23
percentage of participants | 89 | 83

2. Primary Outcome: Percentage of Tetanus Diphtheria Toxoid (Td) Responders at Day 28 Post-Vaccination
Description: Tetanus responders were defined as participants who had at least a 2-fold increase over pre-immunization levels of anti-tetanus antibodies in their blood at 28 days after they were immunized with tetanus.
Time Frame: 28 days after immunization (Day 28 for Vaccinations Only Group/Day 196 for Tysabri Plus Vaccinations Group)
Population: Participants with an assessment at Day 28 and a pre-immunization antibody value ≤ 3.5 IU/mL. No imputation methods were used in the primary analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Tysabri Plus Vaccinations | Vaccinations Only
Number analyzed (Participants) | 16 | 24
percentage of participants | 94 | 100

3. Secondary Outcome: Mean Percentage Change From Baseline in Circulating Lymphocyte Subsets CD3+, CD4+, CD8+, CD19+, and CD56+ at Month 3 of Tysabri Therapy
Description: The effect of Tysabri on circulating lymphocyte subsets (CD3+, CD4+, CD8+, CD19+, and CD56+) was calculated as a percentage change from baseline pre-treatment values (based on absolute count).
Time Frame: Month 0 (Baseline), Month 3
Population: Participants who had received at least 3 doses of Tysabri per protocol; those with insufficient Tysabri dosing or protocol violations were excluded from the relevant analysis population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tysabri Plus Vaccinations
Number analyzed (Participants) | 23
percent change
  CD3+ | 39.6 (26.84)
  CD4+ | 35.7 (26.83)
  CD8+ | 51.8 (36.68)
  CD16+/CD56+ | 68.7 (79.83)
  CD19+ | 135.2 (82.80)

4. Secondary Outcome: Mean Percentage Change From Baseline in Circulating Lymphocyte Subsets CD3+, CD4+, CD8+, CD19+, and CD56+ at Month 6 of Tysabri Therapy
Description: as for outcome 3
Time Frame: Month 0 (Baseline), Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tysabri Plus Vaccinations
Number analyzed (Participants) | 20
percent change
  CD3+ | 52.4 (34.19)
  CD4+ | 48.2 (32.71)
  CD8+ | 67.1 (42.41)
  CD16+/CD56+ | 73.5 (73.20)
  CD19+ | 164.8 (85.21)

5. Secondary Outcome: Mean Alpha4-Integrin Saturation at Baseline, Month 3, and Month 6
Description: Measurement of the degree of natalizumab saturation of the alpha4 integrin on peripheral blood mononuclear cells was accomplished by staining cells with phycoerythrin conjugated anti human IgG4 antibody (hIgG4-PE) to label the cell-bound natalizumab, followed by flow cytometric detection and quantification.
Time Frame: Month 0 (Baseline), Month 3, and Month 6
Population: Participants who received at least 1 dose of Tysabri and had at least 1 post-baseline assessment. n=number of participants with measurement at given timepoint.
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Tysabri Plus Vaccinations
Number analyzed (Participants) | 30
percent saturation
  Baseline; n=27 | 9.9 (16.72)
  Month 3; n=28 | 72.7 (28.93)
  Month 6; n=24 | 80.5 (24.46)

6. Secondary Outcome: Mean Alpha4-Integrin Expression at Baseline, Month 3, and Month 6
Description: Alpha4-integrin expression is the mean fluorescent intensity (MFI), a measure of fluorescence intensity often used to monitor changes in surface antigen modulation in flow cytometry. There is no reference range for this test, which was developed at Biogen Idec.
Time Frame: Month 0 (Baseline), Month 3, and Month 6
Population: Participants who had received at least 1 dose of Tysabri and had at least 1 post-baseline assessment. n=number of participants with measurement at given timepoint.
Measure: Mean (Standard Deviation); unit: mean fluorescent intensity (MFI)
Arm/Group | Tysabri Plus Vaccinations
Number analyzed (Participants) | 30
mean fluorescent intensity (MFI)
  Baseline; n=27 | 633.7 (139.73)
  Month 3; n=28 | 419.5 (158.95)
  Month 6; n=24 | 434.3 (167.93)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from dosing at the Baseline Visit (Month 0) until the participant's End of Study Visit (Month 8). Serious adverse events were collected from screening until 12 weeks following the participant's last dose of Tysabri.
Description: Data for the Tysabri Plus Vaccinations group covers the entire study period, and data for the Vaccines Only group covers only the immunization period.
Groups:
- Tysabri Plus Vaccinations: Participants received 9 monthly doses of Tysabri 300 mg intravenous (IV), and received vaccinations with neoantigen and recall antigen (keyhole limpet hemocyanin [KLH] and tetanus diphtheria toxoid [Td], according to manufacturer's prescribing information) at specified timepoints following the 7th dose.
- Vaccinations Only: Participants received only vaccinations with neoantigen and recall antigen (KLH and Td, according to manufacturer's prescribing information) at specified timepoints. They did not receive any treatment for their MS.
Arm/Group | Tysabri Plus Vaccinations | Vaccinations Only
Serious Adverse Events (participants affected / at risk) | 3/30 | 2/30
Other Adverse Events (participants affected / at risk) | 25/30 | 19/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tysabri Plus Vaccinations (N=30) | Vaccinations Only (N=30)
multiple sclerosis relapse (Nervous system disorders) | 0 | 1
herpes zoster disseminated (Infections and infestations) | 1 | 0
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
angina unstable (Cardiac disorders) | 0 | 1
gastroenteritis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tysabri Plus Vaccinations (N=30) | Vaccinations Only (N=30)
influenza (Infections and infestations) | 4 | 0
bronchitis (Infections and infestations) | 3 | 1
vomiting (Gastrointestinal disorders) | 2 | 0
pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
vision blurred (Eye disorders) | 3 | 0
nasopharyngitis (Infections and infestations) | 2 | 1
fatigue (General disorders) | 3 | 2
diarrhoea (Gastrointestinal disorders) | 2 | 0
oral herpes (Infections and infestations) | 2 | 0
injection site erythrema (General disorders) | 4 | 5
injection site pain (General disorders) | 1 | 7
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
injection site swelling (General disorders) | 0 | 2
paraesthesia (Nervous system disorders) | 4 | 0
injection site warmth (General disorders) | 1 | 2
urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
sinusitis (Infections and infestations) | 3 | 0
pyrexia (General disorders) | 2 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
hypoaesthesia (Nervous system disorders) | 2 | 1
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
upper respiratory tract infection (Infections and infestations) | 2 | 0
urinary tract infection (Infections and infestations) | 3 | 1
otitis media (Infections and infestations) | 2 | 0
fall (Injury, poisoning and procedural complications) | 2 | 0
depression (Psychiatric disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 3 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
multiple sclerosis relapse (Nervous system disorders) | 5 | 5
headache (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.